CLINICAL TRIAL: NCT06149312
Title: A Prospective, Randomized Trial Assessing the Feasibility of an Advance Care Planning Intervention for Patients Hospitalized in a French Cancer Center
Brief Title: Feasibility of an Advance Care Planning Intervention
Acronym: PREVOIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-018; 2023-A02045-40 (Other: ID-RCB Number)
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance Care Planning Intervention (Experimental): Patients from experimental arm will benefit from a Standardized Advance Care Planning interview alone or in the presence of relatives within 3 days after randomization.
  Interventions: Other: Advance Care Planning Intervention
- Standard cares (No Intervention): Patients from control arm will be treated without specific intervention, which does not exclude the possibility of resorting to non standardized advance care planning interviews with an oncologist or a physician specialized in palliative care.

INTERVENTIONS:
Other: Advance Care Planning Intervention — Standardized interview based on The letter Project (Stanford Medicine) and Questions Prompt List
  Arms: Advance Care Planning Intervention

SUMMARY:
Advanced Cancer patients hospitalized in a Cancer center inpatient unit have a dismal prognosis. Palliative Care interventions have shown multiple benefit for those patients, regarding quality of life, symptom management, illness understanding and aggressiveness of care criteria. Although Advance Care planning (ACP) is part of usual Palliative Care, specific interventions dedicated to ACP are understudied.

This study aims at showing that a simple and systematic Advance Care Planning intervention is likely to clarify the understanding of the goals of care by patients, to help with ACP documentation and and potentially to modify the trajectory of illness for patients during and after hospitalization.

DETAILED DESCRIPTION:
PREVOIR is a randomized, single-center, two-arm trial: patients from experimental arm will benefit from a systematic interview on the care plan whereas patients from control arm will received standard cares.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients with a diagnosis of advanced or metastatic solid cancer
* Patients hospitalized in a conventional oncology, radiotherapy or hematology department
* Agreement obtained from the referring oncologist or senior doctor responsible for the patient during hospitalization
* Patient hospitalized for less than 7 days
* Patients who have not yet written advance directives
* Signature of informed consent

Exclusion Criteria:

* Patients treated for hematologic malignancies
* Presence of uncontrolled symptoms that do not allow an interview to be carried out
* Patients with planned hospitalization for chemotherapy or biopsy or performance of a procedure
* Patients < 18 years old or patients ≥ 18 years old under supervision
* Patients placed under judicial protection or guardianship
* Decompensated neuropsychiatric disorders
* Comprehension problems
* Patients without social security
* Allophone patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who write advance directives of living at 3 months | At 3 months from randomization

SECONDARY OUTCOMES:
Percentage of patients who write advance directives of living at 1 month | At 1 month from randomization
Percentage of patients who write advance directives of living at 6 months | At 6 months from randomization
Overall survival | Up to 6 months
Received anti-cancer treatment | up to 6 months
  Prevalence of antineoplastic treatment received within the 3 months that precede death
Patients living trajectory | up to 6 months
  Recording of patient site of death, if applicable

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouleuc C, Savignoni A, Chevrier M, Renault-Tessier E, Burnod A, Chvetzoff G, Poulain P, Copel L, Cottu P, Pierga JY, Bredart A, Dolbeault S. A Question Prompt List for Advanced Cancer Patients Promoting Advance Care Planning: A French Randomized Trial. J Pain Symptom Manage. 2021 Feb;61(2):331-341.e8. doi: 10.1016/j.jpainsymman.2020.07.026. Epub 2020 Jul 31. PMID 32739563